CLINICAL TRIAL: NCT05260801
Title: The Impact of Daytime Light Intensity in Home Workplaces on Health and Well-being of Remote Workers.
Brief Title: The Impact of Light Intensity in Home Workplaces on Remote Workers' Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not receive funding.
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Nina Sharp, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Study 2; NCT04900025 (obsolete NCT alias)
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Daytime Cognitive Performance; Sleep; Alertness
Keywords: Light intensity; Remote workers; Sleep; Cognition

STUDY DESIGN:
Intervention Model Description: Investigators will examine a series of participants (N=36), each of whom will participate in a five-week experiment. Each participant will have a screening visit at their home. The study will be conducted over five successive one-week periods with two cohorts of participants experiencing the same series of lighting interventions. All data collection will be performed during the working days (Monday - Friday) when participants are exposed to the lighting in their home offices.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright lighting followed by Placebo lighting (Experimental): Each lighting condition will last for two weeks (Weeks 2-3 or 4-5), be limited to the 10 workdays, and be active for 8 hours per day. The order of conditions will be randomized.
  Interventions: Other: Bright Lighting; Other: Placebo Lighting
- Placebo lighting followed by bright lighting (Experimental): Each lighting condition will last for two weeks (Weeks 2-3 or 4-5), be limited to the 10 workdays, and be active for 8 hours per day. The order of conditions will be randomized.
  Interventions: Other: Bright Lighting; Other: Placebo Lighting

INTERVENTIONS:
Other: Bright Lighting — The bright lighting condition will administer the light intensity as determined from the finding of Study 1. Bright lighting condition will last for two weeks (Weeks 2-3 or 4-5), be limited to the 10 workdays, and be active for 8 hours per day.
Other: Placebo Lighting — The placebo condition will expose participants to 150 lux, a light level that is equivalent to average room lighting. Placebo lighting condition will last for two weeks (Weeks 2-3 or 4-5), be limited to the 10 workdays, and be active for 8 hours per day. The placebo lighting condition will be applied to minimize the bias and false improvements that might occur due to experiencing new lighting conditions and devices.

SUMMARY:
The lockdowns and restrictions associated with the COVID-19 have created a seismic shift in where work is done. Prior to the pandemic, approximately 20% of individuals were working from home while during the pandemic, more than 70% of individuals worked from home. While it is unlikely that such a large percent of the population will remain working from home, the vast support from workers for such work arrangements and the potential increase in productivity means that there will likely be a revision of the work place with more individuals working from a home office environment than have done so in the past. One unintended aspect of working from home is a reduction in light exposure, especially in the contrast between the daytime and evening. Offices converted from bedrooms, basements, and kitchens are often illuminated in the recommended 50-100 lux range, as opposed to the approximately 500 lux of most offices. While this light intensity is sufficient to work or read by, it may be insufficient to maintain adequate mental and physical health. In addition to light allowing us to consciously perceive the world around us, light can also induce a variety of changes in physiology that can impact our health, notably inducing shifts in the timing of circadian rhythms, suppressing the onset of melatonin production, and increasing alertness with subsequent changes to sleep latency and architecture. These changes in sleep and circadian rhythms have been associated with a variety of pathologies including increased risk of metabolic, psychiatric, cognitive, and cardiovascular disorders, in addition to overall longevity. Development of an adequate prophylactic countermeasure for the circadian desynchrony to which home office workers are exposed is a critical step in maintaining the health of these individuals. There are two main studies. The first study (Years 1-2) will be an in-laboratory determination of the threshold of light needed to minimize the negative impact of nocturnal light exposure. The second study (Years 3-4) will be a field study applying this threshold to determine if whether in situ use of this light intensity during the day improves health and safety among home office workers.

Current CT.gov represents the second part of this study i.e. "Study 2: The impact of daytime light intensity in home workplaces on health and well-being of remote workers. In study 2, investigators will examine a series of participants (N=36), each of whom will participate in a five-week experiment. Each participant will have a screening visit at their home. The study will be conducted over five successive one-week periods with two cohorts of participants experiencing the same series of lighting interventions. All data collection will be performed during the working days (Monday - Friday) when participants are exposed to the lighting in their home offices.

ELIGIBILITY:
Inclusion Criteria:

* Have an occupation of a dayshift (i.e., occurring between 6 AM and 8 PM) remote office worker, working from home for five days (Monday→Friday) a week with a maximum of 12 hours per day.
* Aged 18-65
* Good health [self-reported medical history]
* Female or male
* No evidence of sleep disorders [PSQI scores >5 are excluded]
* No extreme chronotypes (extreme owl or lark) [reduced MEQ scores >27 or <11 are excluded; typical bedtime between 8 PM and 2 AM]
* Non-smoker
* Not abusing alcohol [AUDIT scores >19 are excluded]
* Not experiencing depression [CES-D scores >27 are excluded]
* Best-corrected visual acuity of 20/200 or higher
* Normal color vision [as per Ishihara's Tests for Colour Deficiency]
* No current or planned use of light therapy or light-altering devices (e.g., blue-blocking and/or tinted glasses and contact lenses)
* No planned upcoming travel during the study participation period
* Not pregnant

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Nocturnal Sleep Duration (in minutes) as measured by actigraphy | 24 hours everyday up to week 5
  Nocturnal Sleep Duration (in minutes) will be measured by Actigraphy. Longer sleep duration corresponds to improved sleep outcomes.
Change in Percent Sleep Efficiency (total sleep time divided by time in bed) measured by actigraphy | 24 hours everyday up to week 5
  Percent Sleep Efficiency measured by actigraphy. Higher percentage corresponds to higher sleep quality.
Change in the minutes of wake after sleep onset measured by actigraphy | Everyday up to week 5]
  The investigators will measure patients total time awake between initial sleep onset and the final morning awakening in minutes.
Change in the Subjective Sleep quality as measured by a single Likert-like question qualitatively | everyday up to 5 weeks
  This is included in the consensus sleep diary and consists of 1 question that is scaled from 1 to 7, with higher score corresponds to poor quality sleep.
Change in working memory as assessed by fractal 2-back score | Once on the last day of week 1, 3, and 5
  Fractal 2-back score is based on number of correct responses. Higher test scores indicates better performance of working memory
Change in working Memory as assessed by Visual Object Learning Task (VOLT) score | Once on the last day of week 1, 3, and 5
  Participants first memorize a set of 3-dimensional Euclidean shapes. During recall, participants are to distinguish between the initial shapes mixed with ten distractor shapes. Score is based on number of correct responses.
Change in median reaction time on Psychomotor Vigilance test | Once on the last day of week 1, 3, and 5
  Psychomotor vigilance test(PVT) measures alertness and vigilant attention and is considered to be the gold standard measure of neurobehavioral effects of circadian misalignment and sleep loss. Shorter median reaction times corresponds to more attentive state.
Change in Balloon Analogue Risk Task (BART) score | Once on the last day of week 1, 3, and 5
  Participants inflate balloons of unknown popping probability to obtain the highest reward. Each pump increases the potential reward. The potential reward is lost if the balloon pops.
  Scores are calculated by adding the number of pumps for unexploded balloons, with higher scores reflecting greater risk-taking. Range varies - explosions are at a random point between 1 and 128 pumps.
Change in subjective alertness as assessed by Stanford Sleepiness Scale (SSS) | Once on the last day of week 1, 3, and 5
  SSS is a s self-reported Likert-type sleepiness scale which assess mental and physical sedation and sleepiness, respectively, at that moment and time. SSS only consists of 1 question that is scaled from 1 to 7, with 7 being a higher or worse score (i.e. more sleepy and sedated)

SECONDARY OUTCOMES:
Change in reaction time on Motor Praxis Task (MPT) | Once on the last day of week 1, 3, and 5
  Participants are to quickly touch ever-shrinking boxes. Each time a new box appears in a different location on the screen. Shorter reaction time corresponds to higher sensory motor speed.
Change in measure of abstraction: score on abstract matching test | Once on the last day of week 1, 3, and 5
  Participants select pairs of shapes that fit with another shape. Higher number of correct responses corresponds to higher measure of abstraction.
Change in the spatial orientation: score on line orientation test | Once on the last day of week 1, 3, and 5
  Participants are shown two lines at different angles, and are to rotate one line incrementally until it is parallel to the other. Higher scores corresponds to better spatial orientation.
Change in complex scanning and visual tracking: score on Digit Symbol Substitution Task (DSST) | Once on the last day of week 1, 3, and 5
  Participants touch the number paired to the symbol that matches the current target symbol. Higher score corresponds to better complex scanning and visual tracking capability.

CONTACTS AND LOCATIONS:
Overall Officials: Nastaran Shishegar, PhD, Principal Investigator — Arizona State University

IPD SHARING:
Plan to Share IPD: No